CLINICAL TRIAL: NCT06889584
Title: Evaluating the Efficacy of a Supplement Combination for Improving Stress and Sleep: A Randomized Placebo-Controlled Clinical Trial
Brief Title: Supplement Combination on Stress and Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Momentous (Unknown)
Responsible Party: Principal Investigator, Shawn M. Arent, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00141237
Record Dates: First submitted 2025-02-27; First posted 2025-03-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy
Keywords: Sleep; Stress; Supplement
MeSH Terms: interventions — Ashwagandha; threonic acid; theanine; Apigenin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, between subjects, double-blind.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AM active, PM active (Experimental)
  Interventions: Combination Product: All Active Supplement Combinations (Ashwagandha, Rhodiola rosea, magnesium threonate, L-theanine, and apigenin))
- AM active, PM placebo (Active Comparator)
  Interventions: Combination Product: AM Active Supplement Combination (Ashwagandha and Rhodiola rosea)
- AM placebo, PM active (Active Comparator)
  Interventions: Combination Product: PM Active Supplement Combination (Magnesium threonate, L-theanine, and apigenin)
- AM placebo, PM placebo (Placebo Comparator)
  Interventions: Other: AM and PM Placebo

INTERVENTIONS:
Combination Product: All Active Supplement Combinations (Ashwagandha, Rhodiola rosea, magnesium threonate, L-theanine, and apigenin)) — Ashwagandha, Rhodiola rosea, magnesium threonate, L-theanine, and apigenin.
  Arms: AM active, PM active
Combination Product: AM Active Supplement Combination (Ashwagandha and Rhodiola rosea) — Ashwagandha and Rhodiola rosea
  Arms: AM active, PM placebo
Combination Product: PM Active Supplement Combination (Magnesium threonate, L-theanine, and apigenin) — Magnesium threonate, L-theanine, and apigenin.
  Arms: AM placebo, PM active
Other: AM and PM Placebo — Placebo AM and PM
  Arms: AM placebo, PM placebo

SUMMARY:
The purpose of this clinical trial is to assess the effects of a supplement combination on measures of sleep quality and stress in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants aged 18 to 50 years (inclusive) at the time of screening with a body mass index of 18.5 to 29.9 kg/m2.
* Willing to give voluntary consent, be able to understand and read the questionnaires, carry out all study-related procedures, communicate effectively with the study staff, and agree to allow any study-related evaluations.
* Participant is physically active: participating in resistance and/or endurance exercise ≥150 min/wk for ≥6 mo.
* Participant will be asked about dietary supplementation use within the past 6 months.

If participant began taking a supplement within the past month, participant will be asked to discontinue supplement use followed by a 2-week washout prior to participation.In all other cases, supplement use will be asked to be maintained throughout the study.

• The participant has an apple device with iOS 16 or greater software.

Exclusion Criteria:

* Have a known sensitivity of allergy to any of the investigational products.
* Participants currently taking any of the investigational products will be excluded.
* Female participants who are lactating, pregnant, or planning to become pregnant during the study.
* Diagnosed with any sleep-related or stress-related disorders.
* Currently taking medication to manage sleep or cortisol levels.
* Participants with controlled or uncontrolled hypertension including stage 1 hypertension (systolic blood pressure ≥129 mmHg and diastolic blood pressure ≥89 mmHg).
* Any other condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2026-02-01 (Actual)

PRIMARY OUTCOMES:
Cohen's Perceived Stress scale | Baseline, Day 7, Day 14, Day 21, Day 28
  To determine changes in perceived stress by way of the Cohen's Perceived Stress scale. The minimum is 0 and max is 40, with higher values meaning more stress.
Positive mood and emotion | Baseline, Day 7, Day 14, Day 21, Day 28
  Assessed by the Positive and Negative Affect Scale. Min values of 0 and max of 50, higher scores indicate more positive moods and emotions.
Negative mood and emotion | Baseline, Day 7, Day 14, Day 21, Day 28
  Assessed by the Positive and Negative Affect Schedule. Min values of 0 and max of 50, higher scores indicate more negative moods and emotions.
Weekly sleep disturbances. | Baseline, Day 7, Day 14, Day 21, Day 28
  Assessed by the Patient Reported Outcome Measures of sleep disturbances. Min values of 8 and max values of 40. Higher scores mean more sleep disturbances.
Weekly sleep impairment | Baseline, Day 7, Day 14, Day 21, Day 28
  Assessed by the Patient Reported Outcome Measures of sleep impairments. Min values of 8 and max values of 40. Higher scores mean more sleep impairments.
Changes in daily psychological stress | Daily for 4-weeks from baseline to Day 28.
  Assessed by the Daily Stress Response Scale. Min 0, max 60 with higher scores indicating higher stress.
Changes in daily physiological stress | Daily for 4-weeks from baseline to Day 28.
  Assessed by Daily Stress Response Scale. Min 0, max 60 with higher scores indicating higher stress.
Changes in subjective sleep quality. | Baseline and Day 28.
  Assessed by the Pittsburgh Sleep Quality Index questionnaire. Min 0 and max 21, higher scores indicate worse sleep quality.
Changes in objective sleep quality. | Daily for 4-weeks from baseline to Day 28.
  Assessed by the Absolute Rest device, higher scores are better.
Changes in sleep efficiency. | Daily for 4-weeks from baseline to Day 28.
  Assessed by the Absolute Rest device, total time asleep divided by time in bed, expressed as a percentage, higher is better.
Changes in sleep latency | Daily for 4-weeks from baseline to Day 28.
  Assessed by the Absolute Rest device, time taken to fall asleep.
Changes in sleep duration | Daily for 4-weeks from baseline to Day 28.
  Assessed by the Absolute Rest device, total sleep time.
Changes in sleep apnea | Daily for 4-weeks from baseline to Day 28.
  Assessed by the Absolute Rest device, values measures by oxygen saturation.

SECONDARY OUTCOMES:
Percent compliance of supplement use | End of Week 2 and Week 3.
  To determine the percent of compliance when taking AM and PM pills. Will be measured by the amount of pills taken / pills prescribed multiplied by 100.

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina Sport Science Lab, Columbia, South Carolina, United States